CLINICAL TRIAL: NCT06968247
Title: Assessing the Feasibility of the Patient-Reported Outcomes Based Model for Community Care of Patients With Axial Spondyloarthritis Via a Type 1 Pilot Hybrid Effectiveness-Implementation Trial Using the RE-AIM Framework
Acronym: PROMise-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-4044; AM/HRT048/2025 (SRDUKAMR25H8) (Other Grant/Funding Number: Singapore Health Services PTE LTD)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMise Model of Care (Experimental): Patients will go for blood tests and be sent PROMs questionnaire prior to planned clinic appointments. The results of the blood tests and questionnaire will be reviewed by a physician. The physician will postpone patient's appointment if the patient is assessed as stable. Any physician-endorsed medication will be sent via a medication delivery service.
  Interventions: Procedure: PROMise Model of Care
- Control (No Intervention): Usual care

INTERVENTIONS:
Procedure: PROMise Model of Care — Patients will go for blood tests and be sent PROMs questionnaire prior to planned clinic appointments. The results of the blood tests and questionnaire will be reviewed by a physician. The physician will postpone patient's appointment if the patient is assessed as stable. Any physician-endorsed medication will be sent via a medication delivery service.
  Arms: PROMise Model of Care

SUMMARY:
The goal of this clinical trial is to facilitate the implementation of PROMs-based care for patients with axial spondyloarthritis.

The main questions it aims to answer are:

* What are the barriers, facilitators and strategies to implement PROMs-based care?
* Can the PROMise algorithm successfully review and postpone appointments of eligible patients?
* How feasible is PROMs-based care in patients with axial spondyloarthritis?

Researchers will implement PROMs-Based care and see if PROMs-Based care is feasible and understand patient's opinions on PROMs-Based care implemented.

Participants will:

* Be randomized to either receive intervention (PROM-based care) or control (usual care). Randomisation means assigning you to one of two groups by chance, like tossing a coin or rolling dice.
* That receive PROMs-based care, will be sent PROMs questionnaires that ask them about their health conditions via SMS at a regular interval of 4 months.
* Have their appointments postponed by 4 months, if the PROMise algorithm with specific thresholds (with overview from the rheumatology care team) assess their condition as stable through their blood test results and PROMs questionnaire.
* Have a cap of 12 months between physician visits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with axial spondyloarthritis according to the 2009 ASAS Classification Criteria of AxSpA
* has been receiving care in Singapore General Hospital for at least 6 months
* aged 21 years and above

Exclusion Criteria:

* Bath Ankylosing Spondylitis Disease Activity Index score of >4

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of outpatient rheumatological appointments in 1 year | 1 Year
  To measure the percentage change in the number of outpatient rheumatological appointments in 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Thurah A, Stengaard-Pedersen K, Axelsen M, Fredberg U, Schougaard LMV, Hjollund NHI, Pfeiffer-Jensen M, Laurberg TB, Tarp U, Lomborg K, Maribo T. Tele-Health Followup Strategy for Tight Control of Disease Activity in Rheumatoid Arthritis: Results of a Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2018 Mar;70(3):353-360. doi: 10.1002/acr.23280. Epub 2018 Jan 23. PMID 28511288
- [Background] Kwan YH, Tan JJ, Phang JK, Fong W, Lim KK, Koh HL, Lui NL, Tan CS, Ostbye T, Thumboo J, Leung YY. Validity and reliability of the Ankylosing Spondylitis Disease Activity Score with C-reactive protein (ASDAS-CRP) and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in patients with axial spondyloarthritis (axSpA) in Singapore. Int J Rheum Dis. 2019 Dec;22(12):2206-2212. doi: 10.1111/1756-185X.13735. Epub 2019 Nov 13. PMID 31721427